CLINICAL TRIAL: NCT01365312
Title: A Prospective, Randomized, Blinded, Placebo-Controlled Trial of Periodic, Brief Ethanol Locks to Prevent Peripherally-Inserted Central Catheter (PICC) Infections in Preterm Infants in the Neonatal Intensive Care Unit
Brief Title: Safety and Efficacy Study of Ethanol Locking to Prevent Central Line Infection in Premature Neonates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator relocated
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Amber Fort, Amber Fort, DO, MPH, MS, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NeonatalELT
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Infection Associated With Catheter; Bacteremia; Sepsis
Keywords: Central line associated infection; PICC associated infection; Neonatal central line associated sepsis; Central line colonization; Ethanol Lock
MeSH Terms: conditions — Catheter-Related Infections; Bacteremia; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ethanol (Experimental): Assigned intervention is a 70% ethanol lock, placed every 72 hours for 15 minutes, for the duration of the PICC line.
  Interventions: Drug: Ethanol lock
- Heparinized saline (Placebo Comparator): Intervention is to place a heparinized saline lock every 72 hours for 15 minutes, for the duration of the line.
  Interventions: Drug: Heparinized saline

INTERVENTIONS:
Drug: Ethanol lock — Placement of 0.5 cc 70% ethanol, every 72 hours, for 15 minutes, into PICC lines randomized to ethanol intervention
  Arms: Ethanol
Drug: Heparinized saline — 0.5 cc heparinized saline to be placed once every 72 hours for 15 minutes, in PICC lines randomized to placebo
  Arms: Heparinized saline

SUMMARY:
Appropriate delivery of adequate nutrition and medications in premature infants often requires central venous access in the form of a special IV called a PICC (peripherally inserted central catheter). While a necessary feature of neonatal intensive care, PICCs pose significant risk: among the most serious of these is infection. One common, successful infection control practice used in older children and adults involves the use of a lock, in which a fluid-filled syringe is attached to the end of an IV when it is not in use in order to prevent and/or treat clotting or infection. The solution is left for some period of time and is then either withdrawn from the line or flushed into the patient. The solution could be saline, antibiotics, other antiseptics, or any combination of these. However in the premature infant, use of antibiotics as a locking compound risks leaving behind organisms resistant to treatment; antiseptics can irritate vessels and cause breakage to sensitive premature skin; saline has neither sterilization nor anti-infective properties. By contrast, ethanol neutralizes or kills most bacteria, viruses, and fungi without the risk of resistance, and because it is not externally applied there is no risk to baby skin. Ethanol-based lock protocols have been used safely and effectively in both adult and pediatric populations without adverse effects, but this has not been tested in premature babies because fluids and medication are delivered continuously: placement of a lock traditionally requires an extended pause (hours or days) in fluid and medication administration.

To overcome these key limitations, a periodic, brief ethanol lock protocol was designed such that both infant exposure and interruptions to fluid and medication delivery would be minimized. The lock is practical, cheap, easy to place, and takes advantage of an existing daily pause during which IV tubing and fluids hooked up to the PICC are changed. The objective of this study is to test the hypothesis that use of a 70% ethanol lock, every 3rd day, for 15 minutes, will safely and effectively reduce PICC infection in our unit.

DETAILED DESCRIPTION:
PICC infection is of particular concern in the NICU because of the need for long term intravenous access in many very-low and the majority of extremely-low birthweight infants, the very populations at highest risk for infection in the first place. Central lines are a mainstay of treatment in these babies because of the need for extended parenteral nutrition, which itself has been associated with blood stream infection, not to mention the increased use of anti-infectives, added hospitalization costs, longer length of stay, and negative impact upon nutrition delivery when infectious complications occur.

Existing infection control practices differ by unit and region, and include hand washing, sterile precautions at insertion and dressing changes, elimination of mandatory scheduled dressing changes, minimizing port access to the extent permitted by clinical care, prophylactic antibiotics, and closed medication systems. Success is variable: there is no standard highly effective, safe approach to infection control, and central line infection remains a leading cause of morbidity and mortality in the NICU.

A standard practice to maintain central line patency when it is not in use is to lock it with a syringe containing a heparinized solution. Locks containing antibiotics have been used to prevent infection of central lines and to treat already-infected lines, but this approach confers risk of development of organisms resistant to treatment. External chlorhexidine-impregnated dressings have been used but can harm premature skin and do not achieve sterilization of the lumen or hub, where most infections originate.

Medical grade ethyl alcohol (ethanol) is a widely used compound with uses as a disinfectant, preservative, antidote to ingested ethylene glycol (anti-freeze), and anti-microbial. The FDA lists no specific approval or indication though it's use is widely recognized. Multiple studies have been conducted in sheep, children and adults, using 0.5-2 mL 70% ethanol locks to successfully prevent and/or treat catheter related infection without development of resistant organisms, adverse side effects to patients, or disruptions in catheter integrity. Though the ethanol lock approach has not yet been applied to premature neonates, safe and successful precedent in humans as young as 3 months is established; ours is the first trial of ethanol locking in a NICU setting.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants < 32 weeks gestation at birth who require a PICC

Exclusion Criteria:

* Any baby with a positive blood culture less than 48 hours prior to PICC placement; any infant who requires pressors in excess of >5 mcg/kg/min

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incidence of PICC-related sepsis in infants with ethanol-treated vs. Placebo treated lines | Study Day #28 or sooner if PICC is discontinued before day #28
  Primary endpoint of the study is to compare the incidence of PICC-related sepsis in infants with ethanol treated vs. Placebo treated lines by study day 28. PICC-related sepsis is defined by any 2 clinical signs or symptoms plus one positive peripheral blood culture for a recognized pathogen in this population other than coagulase-negative staphylococcus, or 2 positive peripheral blood cultures for coagulase-negative staphylococcus within 48 hours.

SECONDARY OUTCOMES:
Evaluation of PICC colonization following ethanol locking | Duration of PICC use, average of 3 weeks
  PICC colonization is reflected by growth of >15 CFU from a 5-cm segement of the PICC tip by semiquantitative (roll-plate) culture, or growoth of >100 CFU by quantitative (sonication) broth culture in an otherwise asymptomatic patient.
Whether the primary and secondary endpoints differ by birthweight strata | Duration of PICC use, average of 3 weeks
  Birthweight stratification will use a 3-tiered subset (<1000g, 1000-1250g, and >1250g) consistent with existing neonatal literature.
To determine whether ethanol lock treatment impacts incidence of clinical evaluations for suspected sepsis | Duration of PICC use, average of 3 weeks
  Other evaluations for suspected sepsis are those not defined by the primary endpoint but meeting criteria for infection of some other sterile body fluid (urine or CSF).
To determine whether antibiotic use for any indication (including non-bacteremia) alters the incidence of PICC-related infection or colonization as defined in the primary and secondary endpoints | Duration of PICC use, average of 3 weeks
  See above
Determine side effects of ethanol locking in premature babies | Duration of PICC use, average of 3 weeks
  To determine the side effects of flushing ethanol locks into premature infants following lock therapy, if any
To determine effect of ethanol locking on neonatal PICC lines | Duration of PICC use, average of 3 weeks
  To determine how ethanol locking affects central line function and integrity in vivo, if at all.

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Greenville, North Carolina, United States